CLINICAL TRIAL: NCT02756000
Title: Appropriate Timing of Complete Revascularization for Multivessel Coronary Artery Disease After Culprit Only Primary Percutaneous Coronary Intervention (PCI) for ST Elevation Myocardial Infarction
Brief Title: Timing of Complete Revascularization for Multivessel Coronary Artery Disease in STEMI
Acronym: MVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center Zemun (Other)
Collaborators: Institute of Cardiovascular Diseases, Vojvodina (Other); Military Medical Academy, Belgrade, Serbia (Other); Clinical Center Kragujevac, Kragujevac, Serbia (Unknown)
Responsible Party: Principal Investigator, Ivan Ilic, Head of interventional cardiology diagnostics, Clinical Hospital Center Zemun
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEM-CARD-003
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; percutaneous coronary intervention; multivessel coronary artery disease; dobutamine stress echocardiography
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- complete PCI at initial hospitalization (Experimental): Staged, complete revascularization of all non-culprit significant lesions in a single PCI session during initial hospitalization for ST elevation myocardial infarction
  Interventions: Procedure: PCI
- complete PCI after 30 days (Experimental): Staged, complete revascularization of all non-culprit significant lesions in a single PCI session after 30 days from initial hospitalization for ST elevation myocardial infarction
  Interventions: Procedure: PCI
- Dobutamine stress testing (Active Comparator): Revascularization by PCI or deferral of revascularization of non-culprit coronary artery lesions based on ischemia testing using Dobutamin stress echocardiography
  Interventions: Procedure: PCI; Procedure: dobutamine stress echocardiography

INTERVENTIONS:
Procedure: PCI — percutaneous angioplasty and stent implantation in coronary artery with significant atherosclerosis and stenosis
  Other Names: percutaneous coronary intervention
Procedure: dobutamine stress echocardiography — Echocardiographic stress test of provoked myocardial ischemia using dobutamine
  Arms: Dobutamine stress testing

SUMMARY:
The study will compare clinical outcomes between complete revascularization during hospitalization for ST elevation myocardial infarction (STEMI) and intervention after 30 days and intervention based on outpatient non-invasive ischemia testing in patients with multivessel coronary artery disease (MVD) presenting with first ever ST elevation myocardial infarction.

DETAILED DESCRIPTION:
This study is prospective, randomized, multicentre, open label study in patients with ST elevation myocardial infarction (STEMI) with multivessel coronary artery disease (MVD) defined as >70% stenosis in a non-culprit vessel, initially treated with culprit only primary PCI. The patients will be enrolled in four high volume PCI centers after successful culprit only primary PCI and then randomly assigned to one of three treatment arms:1. complete revascularization of all non-culprit significant lesions in a single session during initial hospitalization; 2. same revascularization in a single session after 30 days; 3.revascularization or it's deferral based on ischemia testing using Dobutamin stress echocardiography. The study will explore differences in occurrence of major adverse cardio-cerebral events (cardiac death, repeated myocardial infarction, cerebrovascular accident and repeated revascularization) and complications of interventions during 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and electrocardiographic signs of first ever ST elevation myocardial infarction (chest pain lasting less than 12 hours with persistent ST elevation of ≥ 1mm in two contiguous leads on ECG recording)
* Multivessel coronary artery disease (MVD) on initial coronary angiogram, defined as visually assessed stenosis of more than 70% of any of the non-culprit vessels
* Treated with primary PCI of infarct related artery (IRA) only.

Exclusion Criteria:

* Hemodynamically unstable patients defined as presence of cardiogenic shock, intraaortic balloon pump (IABP) implantation and mechanical ventilation prior, during and after primary PCI;
* Presence of significant valvular disease;
* Decision that patient needs to be treated with coronary artery bypass graft (CABG) and/or valvular replacement or reconstruction surgery after initial culprit only PCI;
* Myocardial infarction is caused by stent thrombosis:
* Chronic total occlusion of any of the coronary arteries on initial angiogram;
* Previously treated by CABG surgery;
* Estimated life expectancy less than one year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
major adverse cardio-cerebral events | one year
  cardiac death, repeated myocardial infarction, cerebrovascular accident and repeated revascularization

SECONDARY OUTCOMES:
cardiac death | one year
  Occurence of death caused by cardiac condition
repeated myocardial infarction | one year
  Occurrence of repeated myocardial infarction in the study groups
complications of percutaneous coronary intervention | one year
  Occurrence of vascular complications of PCI, contrast induced nephropathy (CIN) and bleeding events
stent thrombosis | two years
  Occurrence of stent thrombosis based on Associated Research Consortium (ARC) criteria
hospitalization for heart failure | one year
  Occurrence of hospitalization for heart failure in the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar N Neskovic, MD, PhD, Study Chair — Clinical Hospital Center Zemun
Locations (4):
- Serbia (4):
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Institute for cardiovascular diseases Vojvodine, Novi Sad

IPD SHARING:
Plan to Share IPD: Undecided